CLINICAL TRIAL: NCT05179694
Title: A Randomised Controlled Trial Comparing TRANSrectal Biopsy Versus Local Anaethetic Transperineal Biopsy in Evaluation (TRANSLATE) of Men With Potential Clinically Significant Prostate Cancer
Brief Title: The TRANSLATE Trial
Acronym: TRANSLATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 15497-SP001-AC001
Record Dates: First submitted 2021-10-14; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-10

CONDITIONS: Prostate Cancer
Keywords: Biopsy; Transrectal biopsy; Local anaesthetic transperineal biopsy; Pathology; Infection; Tolerability; Complications; Health economics
MeSH Terms: conditions — Prostatic Neoplasms; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local Anaesthetic Transperineal Prostate Biopsy (LATP) (Experimental): LATP prostate biopsy performed with an average of 12 biopsy cores in 6 sectors depending on prostate size, plus typically 4 target cores per MRI lesion, using an ultrasound probe-mounted LATP needle guidance device (e.g. the "Precision-Point" access system, or BK UA1232, or any other which is used in a virtually identical fashion).
  Interventions: Diagnostic Test: Prostate biopsy
- Transrrectal Ultrasound-guided Prostate Biopsy (TRUS) (Active Comparator): TRUS prostate biopsy performed according to each hospital's standard practice, with an average of 12 biopsy cores, in two sectors with additional target pots (typically 4 target cores per MRI lesion).
  Interventions: Diagnostic Test: Prostate biopsy

INTERVENTIONS:
Diagnostic Test: Prostate biopsy — Prostate biopsy via either the Transrectal route (comparator) or Transperineal route (experimental), each under local anaesthetic.

SUMMARY:
The TRANSLATE randomised controlled trial aims to evaluate local anaesthetic transperineal biopsy (LATP) versus transrectal ultrasound-guided (TRUS) prostate biopsy, in the evaluation of previously biopsy-naive men being investigated for clinically significant prostate cancer (on the basis of an elevated age-specific PSA, or abnormal digital rectal examination, or MRI-visible lesion). Men under investigation for possible prostate cancer and recruited to TRANSLATE will be randomised to receive either an LATP or TRUS prostate biopsy, with the primary outcome measure being detection of clinically significant prostate cancer (defined as any Gleason pattern 4 disease, i.e. any Gleason Grade Group >=2 disease). Secondary outcome measures include infection, other complications, tolerability, rate of re-biopsy, detection of clinically insignificant prostate cancer, and a full health economics evaluation.

DETAILED DESCRIPTION:
100,000 men each year in the United Kingdom are referred for investigation for possible prostate cancer based on an abnormal digital rectal examination of the prostate and/or an elevated age-specific PSA blood test. These men may be offered a pre-biopsy MRI scan, followed by a prostate biopsy. Prostate biopsies have typically been taken via an ultrasound-guided transrectal approach (TRUS) under local anaesthetic in the clinic for several decades. However, local anaesthetic transperineal biopsy (LATP) has been pioneered in recent years, in order to sample the prostate gland via the perineum in the clinic, with the potential advantage that the transperineal approach to sampling reduces the risk of serious infection, and improves the sampling of the prostate gland (thus increasing the cancer detection), whilst avoiding the need for general anaesthetic in the operating theatre (as was the case for historical template prostate biopsies).

The way in which urologists take biopsies for possible prostate has started to vary across the United Kingdom; however, no level 1 evidence exists as to which method is best - both in terms of detecting clinically significant prostate cancer, and in terms of the occurrence of serious infection and other common side-effects of the biopsy process, along with patient tolerability, re-biopsy rate, and cost-effectiveness.

The TRANSLATE study aims to recruit 1042 men from at least 9 large Urology departments from United Kingdom Hospitals. These men will be under investigation for possible prostate cancer, and will not have received a prostate biopsy previously.

All men eligible for the study will have had a pre-biopsy MRI scan as part of the investigation for possible prostate cancer. After obtaining informed consent they will be randomised to either a TRUS biopsy or an LATP biopsy. Following the biopsy procedure, the study team will follow up the men in order to determine the rate of detection of clinically significant prostate cancer (primary outcome) in each biopsy group. The study team will also gather information (as secondary outcomes) on the occurrence of any post biopsy infections, and other patient reported biopsy-related complications such as bleeding, bruising, pain, and loss of erections and sexual function. Additionally, the study team will record any subsequent prostate biopsy procedures, which might be recommended if the first prostate biopsy has produced a possible 'false negative' result, where clinicians have concerns that the prostate biopsy result is inconsistent with the pre-biopsy MRI scan result and where there are concerns that a 'clinically significant' prostate cancer may have been under-detected. Data will be collected before the biopsy (baseline), immediately after the biopsy, and then at 7 days, 35 days and 4 months following the biopsy.

The total length of the study is 31 months (to include trial setup phase, recruitment phase, data analysis and write-up of reports and publications). Recruitment of patients will last for 15 months. There will be a formal 'stop/go' review at the end of month 12 (i.e. after a full 6 months of recruitment) in order to ensure that a minimum of 140 patients has been randomised, and that at least 4 centres have been opened to recruitment. If the study team meets the 'stop/go' recruitment target, the trial will continue to recruit for a further 9 months. Data from all patients recruited in the 15 month period will be included in the final analysis.

ELIGIBILITY:
Inclusion Criteria:

All biopsy-naïve men aged 18 years and over who, during investigation for suspicion of possible prostate cancer, require a prostate biopsy. This includes:

* A PSA value above the age-adjusted upper limit of normal, regardless of the MRI result, OR An abnormal pre-biopsy MRI on a 1.5 Tesla or higher MRI scanner, OR An abnormal prostate DRE (regardless of serum PSA or MRI result)
* Considered suitable to tolerate an LATP biopsy procedure by the local clinical team
* Able to give informed consent
* Able to understand written English to enable completion of study validated patient reported outcome measures (questionnaires).

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* Any previous prostate biopsy
* Dysuria on the day of biopsy or untreated urinary tract infection (UTI)
* Immunocompromised (due to history of prior immunocompromising medical condition, or medications e.g. steroids or methotrexate)
* May need enhanced antibiotic prophylaxis: Indwelling catheter, recurrent UTIs
* Previous abdomino-perineal resection (i.e. absent rectum)
* Unable to recline adequately in Lloyd-Davis / lithotomy position (e.g. hip surgery, contractures)
* Unable to have a pre-biopsy MRI (e.g. pacemaker, eGFR <50, claustrophobia)
* PSA >50 ng/ml (i.e. locally advanced/metastatic prostate cancer easily detectable by TRUS).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1042 (Estimated)
Dates: Start 2021-12-03 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Detection of clinically significant prostate cancer. | 4 weeks
  Clinically significant prostate cancer (as defined by the presence of Gleason Grade Group ≥2 prostate cancer, i.e. any Gleason pattern ≥4 disease).

SECONDARY OUTCOMES:
Infection | 7 days, 35 days, and 4 months post procedure.
  Post-biopsy infection - patient questionnaire reporting.
Health-related quality of life. | At baseline, 7 days, 35 days and 4 months post procedure.
  Patient reporting.
Patient reported tolerability of the procedure. | Immediately post-procedure.
  ProBE questionnaire.
Patient reported biopsy-related complications. | 7 days post-procedure.
  ProBE questionnaire.
Number of subsequent prostate biopsy procedures required. | 7 days, 35 days, and 4 months post procedure.
  Patient reporting.
Cost-effectiveness. | Baseline, 7 days, 35 days and 4 months post procedure.
  Resource use questionnaire.
Histological parameters (ISUP grade group, cancer core length, core involvement, target biopsy cancer parameters). | Within 4 weeks of biopsy.
  Histology reporting of grading of biopsy samples as per local reporting practices.
Serious adverse events incidence. | Up to 4 months post procedure.
  Patient questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bryant, Principal Investigator — University of Oxford; Alastair Lamb, Principal Investigator — University of Oxford
Locations (1):
- Department of Urology, Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bryant RJ, Marian IR, Williams R, Lopez JF, Mercader C, Raslan M, Berridge C, Whitburn J, Campbell T, Tuck S, Barber VS, Scaife J, Hewitt A, Taylor A, Ooms A, Landeiro F, Little M, Wolstenholme J, Ghosh S, Reynard JM, Hamdy FC, Liew MPC, Leslie TA, Catto JWF, Rosario DJ, Omer A, Good DW, Gray RH, Kommu S, Chung D, Wells H, Narahari K, Macpherson RE, Verrill C, Eddy B, Yamamoto H, Lamb AD; TRANSLATE Trial Study Group. Local anaesthetic transperineal biopsy versus transrectal prostate biopsy in prostate cancer detection (TRANSLATE): a multicentre, randomised, controlled trial. Lancet Oncol. 2025 May;26(5):583-595. doi: 10.1016/S1470-2045(25)00100-7. Epub 2025 Mar 23. PMID 40139210
- [Derived] Marian IR, Ooms A, Holmes J, Parkes MJ, Lamb AD, Bryant RJ. Statistical analysis plan for the TRANSLATE (TRANSrectal biopsy versus Local Anaesthetic Transperineal biopsy Evaluation of potentially clinically significant prostate cancer) multicentre randomised controlled trial. Trials. 2024 Jun 14;25(1):383. doi: 10.1186/s13063-024-08224-4. PMID 38872174
- [Derived] Kaplan-Marans E, Zhang TR, Hu JC. Differing Recommendations on Prostate Biopsy Approach to Minimize Infections: An Examination of the European Association of Urology and American Urological Association Guidelines. Eur Urol. 2023 Nov;84(5):445-446. doi: 10.1016/j.eururo.2023.05.036. Epub 2023 Jun 7. PMID 37296040